CLINICAL TRIAL: NCT02853604
Title: Phase 3 Study of ADXS11-001 Administered Following Chemoradiation as Adjuvant Treatment for High Risk Locally Advanced Cervical Cancer: AIM2CERV
Brief Title: Study of ADXS11-001 in Participants With High Risk Locally Advanced Cervical Cancer
Acronym: AIM2CERV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADXS001-02; 2015-004844-20 (EudraCT Number)
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: High Risk Cervical Cancer; Advanced Cervical Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants with locally advanced cervical cancer at higher risk for recurrence (HRLACC) received ADXS11-001 matching placebo by intravenous infusion for approximately 60 minutes every 3 weeks for 3 doses (Weeks 1, 4 and 7) and thereafter, every 8 weeks for 5 doses (Weeks 15, 23, 31, 39, and 47) during treatment phase or until disease recurrence. Participants received a 7-day course placebo matching to either trimethoprim/sulfamethoxazole or ampicillin starting 72 hours post treatment in prime and maintenance phase.
  Interventions: Drug: Placebo
- ADXS11-001 (Experimental): Participants with HRLACC received ADXS11-001 at a dose of 1x10^9 colony forming units (CFU) by intravenous infusion for approximately 60 minutes every 3 weeks for 3 doses (Weeks 1, 4 and 7) and thereafter, every 8 weeks for 5 doses (Weeks 15, 23, 31, 39, and 47) during treatment phase or until disease recurrence. Participants received a 7-day course of either trimethoprim/sulfamethoxazole or ampicillin starting 72 hours post treatment in prime and maintenance phase.
  Interventions: Drug: ADXS11-001

INTERVENTIONS:
Drug: ADXS11-001
  Arms: ADXS11-001
Drug: Placebo
  Arms: Placebo

SUMMARY:
Locally advanced cervical cancer at higher risk for recurrence (HRLACC) following concurrent chemotherapy and radiation therapy. This is a group of participants with a significant unmet need. The estimated probability of disease recurrence or death within 4 years of diagnosis is 50% and the prognosis is very grave for those who experience a recurrence.

The purpose of the study was to compare the disease free survival (DFS) of ADXS11-001 to placebo administered following cisplatin-based combination chemotherapy and radiation (CCRT) with curative intent in participants with HRLACC.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled randomized study of ADXS11-001 administered in the adjuvant setting after completion of CCRT in participants with HRLACC, or death. All eligible participants had received CCRT administered with curative intent according to institutional/national guidelines as well as meeting the minimum standards defined in the protocol. Participants initiated the Screening period within 10 weeks after the completion of CCRT. Baseline radiographic assessments and clinical laboratory assessments were completed no longer than 28 days prior to and 3 days prior to the first study treatment infusion, respectively. Eligible participants were randomized 1:2 to receive either placebo or ADXS11-001. Participants received 1 infusion of study treatment administered every 3 weeks for 3 doses for the first 3 months. Thereafter, participants received study treatment every 8 weeks for a total of 5 doses or until disease recurrence. Participants received a 7-day course of an oral antibiotic or placebo starting 72 hours following the completion of study treatment administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a biopsy confirmed diagnosis of squamous cell, adenocarcinoma, or adenosquamous carcinoma of the cervix. Histologic confirmation of the original primary tumor is required.
* Participants with HRLACC.
* Participants included those with stage IB2, IIA2, IIB with pelvic lymph node metastases; all FIGO Stage IIIA, IIIB, IVA or any FIGO Stage (except stage IVB) with para-aortic lymph node metastases as defined by the FIGO 2014 staging criteria for carcinoma of the cervix uteri.
* Participants must have received definitive therapy with curative intent, which consist of at least 4 weeks of treatment with cisplatin and a minimum of 40Gy external beam radiation therapy (EBRT).
* Have performance status of 0 or 1 on the gynaecologic Oncology Group (GOG) performance scale
* Demonstrate adequate organ function

Exclusion Criteria:

* Has not achieved disease-free status after completion of CCRT administered with curative intent.
* Has International Federation of Gynecology and Obstetrics (FIGO) Stage IVB
* Has histologies other than squamous cell, adenocarcinoma, or adenosquamous carcinoma of the cervix.
* Has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)).
* Has a contraindication (sensitivity or allergy) to trimethoprim/sulfamethoxazole and ampicillin.
* Has undergone a previous hysterectomy defined as removal of the entire uterus or will have a hysterectomy as part of their initial cervical cancer therapy. NOTE: Women who have had a partial/subtotal hysterectomy are eligible to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (41):
  - Mobile, Alabama
  - Site, Phoenix, Arizona
  - Phoenix, Arizona
  - Duarte, California
  - Long Beach, California
  - Site, Orange, California
  - Orange, California
  - Site, San Francisco, California
  - Site, Miami, Florida
  - Site, Tallahassee, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Maywood, Illinois
  - Site, Park Ridge, Illinois
  - Site, Indianapolis, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Scarborough, Maine
  - Site, Baltimore, Maryland
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Site, Omaha, Nebraska
  - Site, Las Vegas, Nevada
  - Site, Hackensack, New Jersey
  - Site, Newark, New Jersey
  - Albany, New York
  - Site, Brooklyn, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Site, Cincinnati, Ohio
  - Site, Hilliard, Ohio
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Site, Dallas, Texas
  - Site, Galveston, Texas
  - Houston, Texas
  - Milwaukee, Wisconsin
- Site, La Rioja, Argentina
- Brazil (2):
  - Site, Rio de Janeiro, Rio de Janeiro
  - Site, Natal, Rio Grande do Norte
- Canada (3):
  - SITE, Calgary, Alberta
  - SITE, Montreal, Quebec
  - Site, Sherbrooke, Quebec
- Chile (2):
  - SITE, Temuco, Región de la Araucanía
  - SITE, Santiago, Santiago Metropolitan
- Malaysia (4):
  - Site, Kota Bharu, Kelantan
  - Site, Ampang, Selangor
  - Site, Kuala Lumpur
  - Site, Pulau Pinang
- Mexico (2):
  - Site, Mexico City, D.F.
  - Site, Chihuahua City
- Poland (2):
  - Site, Bialystok
  - Site, Lublin
- Russia (13):
  - Site, Krasnodar, Krasnodarskiy Kray
  - Site, Arkhangelsk
  - Site, Moscow
  - Site, Nal'chik
  - Site, Nizhny Novgorod
  - Site, Obninsk
  - Site, Orenburg
  - Site, Pyatigorsk
  - Site, Rostov-on-Don
  - Site, Saint Petersburg
  - Site, Sochi
  - Site, Ufa
  - Site, Volgograd
- Serbia (3):
  - Site, Belgrade
  - Site, Kamenitz
  - Site, Kragujevac
- South Korea (3):
  - Site, Seongnam
  - Site, Seoul
  - Site, Yangsan
- Spain (12):
  - Site, Barcelona
  - Site, Córdoba
  - Site, El Palmar
  - Site, Elche
  - Site, Girona
  - Site, Madrid
  - Site, Málaga
  - Site, Palma de Mallorca
  - Site, Sabadell
  - Site, Seville
  - Site, Valencia
  - Site, Zaragoza
- Taiwan (4):
  - Site, Taichung
  - Site, Tainan
  - Site, Taipei
  - Site, Taoyuan District
- Ukraine (10):
  - Site, Chernivtsi
  - Site, Dnipro
  - Site, Ivano-Frankivsk
  - Site, Kharkiv
  - Site, Khmelnytskyi
  - Site, Lutsk
  - Site, Poltava
  - Site, Ternopil
  - Site, Vinnytsia
  - Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander LM, van Pijkeren JP. Modes of therapeutic delivery in synthetic microbiology. Trends Microbiol. 2023 Feb;31(2):197-211. doi: 10.1016/j.tim.2022.09.003. Epub 2022 Oct 8. PMID 36220750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with high-risk disease as determined by prognostic factors such as tumor staging, nodal involvement, extent of nodal involvement, and location of nodal involvement were enrolled in this study.
Pre-assignment Details: Participants completed cisplatin-based combination chemotherapy and radiation (CCRT) before enrollment into the study.
Period: Overall Study
Arm/Group | Placebo | ADXS11-001
Started | 37 | 73
Treated | 37 | 72
Completed | 9 | 21
Not Completed | 28 | 52
Not completed — Withdrawal by Subject | 12 | 35
Not completed — Lost to Follow-up | 4 | 8
Not completed — Death | 1 | 5
Not completed — Miscellaneous | 11 | 2
Not completed — Progressive Disease | 0 | 2

BASELINE CHARACTERISTICS:
Population: The As Treated (AT) Population included all participants who received any dose of the study treatment.
Groups:
- Placebo: Participants with HRLACC received ADXS11-001 matching placebo by intravenous infusion for approximately 60 minutes every 3 weeks for 3 doses (Weeks 1, 4 and 7) and thereafter, every 8 weeks for 5 doses (Weeks 15, 23, 31, 39, and 47) during treatment phase or until disease recurrence. Participants received a 7-day course placebo matching to either trimethoprim/sulfamethoxazole or ampicillin starting 72 hours post treatment in prime and maintenance phase.
- ADXS11-001: Participants with HRLACC received ADXS11-001 at a dose of 1x10^9 CFU by intravenous infusion for approximately 60 minutes every 3 weeks for 3 doses (Weeks 1, 4 and 7) and thereafter, every 8 weeks for 5 doses (Weeks 15, 23, 31, 39, and 47) during treatment phase or until disease recurrence. Participants received a 7-day course of either trimethoprim/sulfamethoxazole or ampicillin starting 72 hours post treatment in prime and maintenance phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | ADXS11-001 | Total
Number analyzed (Participants) | 37 | 72 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (10.34) | 49.3 (10.61) | 48.2 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 72 | 109
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 15 | 23
  Not Hispanic or Latino | 28 | 57 | 85
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 30 | 53 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS was defined as the time from randomization until death or recurrence. The date of recurrence was defined as the date of the first time point when recurrence of disease was determined. The determination of recurrence should occur by definitive pathologic tissue confirmation (e.g., biopsy/fine needle aspirate). However, in those cases where it was not medically feasible to obtain a tissue sample then radiographic evidence, when confirmed by independent radiology review, was used to determine recurrence.
Time Frame: From the time of randomization to recurrence or death (Maximum duration: 44.7 months)
Population: This endpoint was not reported as the study was terminated early due to business reasons, therefore, no efficacy data was collected.
Arm/Group | Placebo | ADXS11-001
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Adverse event (AE): any untoward medical occurrence in a participant administered a study treatment & which did not necessarily have to have a causal relationship with the study treatment. An AE is, any unfavorable & unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of study treatment. AE with onset dates on or after the first dose of study treatment were considered treatment emergent.
Time Frame: From first dose of study drug until end of study (Up to 44.7 months)
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ADXS11-001
Number analyzed (Participants) | 37 | 72
Participants | 30 | 62

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization until death due to any cause.
Time Frame: From the date of randomization until death due to any cause (Maximum duration: 44.7 months)
Population: as for outcome 1
Arm/Group | Placebo | ADXS11-001
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study (Up to 44.7 months)
Description: AT Population
Groups:
- Placebo: Participants with HRLACC received ADXS11-001 matching placebo by intravenous infusion for approximately 60 minutes every 3 weeks for 3 doses (Weeks 1, 4 and 7) and thereafter, every 8 weeks for 5 doses (Weeks 15, 23, 31, 39, and 47) during treatment phase until or disease recurrence. Participants received a 7-day course placebo matching to either trimethoprim/sulfamethoxazole or ampicillin starting 72 hours post treatment in prime and maintenance phase.
Arm/Group | Placebo | ADXS11-001
All-Cause Mortality (participants affected / at risk) | 1/37 | 5/72
Serious Adverse Events (participants affected / at risk) | 3/37 | 10/72
Other Adverse Events (participants affected / at risk) | 30/37 | 62/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | ADXS11-001 (N=72)
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | ADXS11-001 (N=72)
Anaemia (Blood and lymphatic system disorders) | 3 | 14
Leukopenia (Blood and lymphatic system disorders) | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3
Monocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 8
Eye irritation (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4
Defaecation urgency (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 20
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 10
Asthenia (General disorders) | 3 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 0 | 23
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 13
Feeling cold (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 11
Influenza like illness (General disorders) | 0 | 3
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 0
Pain (General disorders) | 2 | 3
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 27
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 11
Acarodermatitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Immune system disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Vaginal infection (Infections and infestations) | 1 | 1
Viral sinusitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Drug administration error (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 2 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 2
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood chloride decreased (Investigations) | 0 | 3
Blood pressure increased (Investigations) | 0 | 2
Blood urea increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 0 | 6
Lymphocyte count decreased (Investigations) | 1 | 2
Mean cell haemoglobin decreased (Investigations) | 0 | 1
Mean cell volume decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 2
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 7 | 20
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 2 | 1
Irritability (Psychiatric disorders) | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Ureteric dilatation (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Cervix inflammation (Reproductive system and breast disorders) | 0 | 1
Coital bleeding (Reproductive system and breast disorders) | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 2 | 2
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Hydrometra (Reproductive system and breast disorders) | 1 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 4
Uterine pain (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 2 | 3
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal adhesion (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 2
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 4
Hypotension (Vascular disorders) | 5 | 14
Pallor (Vascular disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall seek the Sponsor's written approval for study results publication which shall not be unreasonably withheld. Such publication by Institution and/or Investigator may be no earlier than after a cooperative publication has been published with Sponsor or 1 year from date of completion or termination of the Study & only after review and comment by Sponsor. Institution agrees to provide Sponsor a copy of proposed publication at least 60 days prior to submission to a publisher.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT02853604/Prot_SAP_000.pdf